CLINICAL TRIAL: NCT05654584
Title: Evaluation of the Relationship Between Weight Loss and Aggression After Laparoscopic Sleeve Gastrectomy Surgery
Brief Title: Weight Loss and Aggression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, Uzman Doktor, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: ANILERGİNNN
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Obesity; Obesity, Morbid; Aggression
Keywords: agression; obesity; laparoscopic sleeve gastrectomy; morbid obesity
MeSH Terms: conditions — Obesity; Obesity, Morbid; Aggression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- agression before surgery: The group that the aggression assessment when morbidly obese before surgery
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- agression after surgery: group reassessed for aggression following postoperative weight loss
  Interventions: Procedure: laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy — Laparoscopic sleeve gastrectomy surgery will be performed by a single surgeon.

SUMMARY:
Obesity has become an important medical and social problem in western countries today. Although many surgical procedures are performed for obesity, Laparoscopic sleeve gastrectomy (LSG) has become the most common bariatric procedure in obesity. The absence of digestive anastomosis, the absence of mesenteric defects that may cause internal hernias and foreign materials such as gastric band are among the advantages of this surgical method.

Obesity is a complex multifactorial disease. Obesity is not a mental disorder, but is associated with serious serious conditions and increases the risk of mental disorders. The social label of obesity will have long-lasting devastating effects on mental health. In addition, obesity is associated with undesirable conditions; Misperception of dietary needs, self-perceived health status and potential social isolation, negative attitude towards appearance, aggression, depression, anxiety, attention deficit/hyperactivity disorder, behavioral problem, and bullying are some of the problems associated with obesity. Body changes are important in the experience of being different from their peers and can result in lowered self-esteem and be a barrier to social functioning. Studies on this condition have shown that obese subjects have poor social functioning and social skills.

There are many factors that cause aggression, but obesity is one of them. Although there are many studies examining the relationship between overweight and aggression in children and adolescent patient groups, studies examining the adult patient group are limited. Starting from this point, we aimed to determine the change in aggression after weight loss in patients who underwent LSG surgery in the study we created.

DETAILED DESCRIPTION:
Fifty patients who underwent laparoscopic sleeve gastrectomy due to morbid obesity in Fatih Sultan Mehmet Training and Research Hospital General Surgery Clinic will be included in the study. The number of samples was calculated by performing impact power analysis. Informed consent form and voluntary consent form will be obtained from all patients.

One month before the surgery, the patients will be weighed and their body mass indexes will be calculated. On the same day, patients will have to fill out the Buss-Perry Aggression Scale questionnaire. LSG operation will be applied to all patients as standard. The patients will be weighed again in the 6th month after the operation, and their body mass indexes will be calculated and recorded. The Buss-Perry Aggression Scale questionnaire will be applied to the patients on the same day. Survey results will be saved in excel. Patients who lost less than 10% of their initial weight for surgery within six months will not be included in the study. Validity and Reliability study of the Turkish version of the Buss-Perry Aggression Scale has been done and it has been mentioned in the sources. Patients will be evaluated in terms of age, gender, BMI (body mass index), comorbidities, marital status and whether they have been diagnosed with depression before.

Standard LSG operating procedure: Five trocar techniques are used and the surgeon stands between the patient's legs. After induction of general anesthesia, the patient is placed in the supine inverted Trendeleburg position and the optiview trocar (Ethicon Endo-surgery, Cincinnati Ohio) is used to enter the peritoneal cavity. LSG begins with the division of the vascular supply of the greater curvature of the stomach, the gastrocolic and gastrosplenic ligaments are cut very close to the stomach. The dissection is continued until the left crus of the diaphragm, the gastrophrenic ligament is divided, the gastric fundus is completely freed, and it is ready to be excised. After this step, a 46 Fr(French) boogie is placed in the stomach and gastrectomy provides a tight tube starting from approximately 5 cm proximal to the pylorus. The procedure continues with a longitudinal gastrectomy of the greater cruciate of the stomach. An Echelon stapler is used with the 60mm Echelon Compact Linear Cutter loaded with ECR60D cartridges (Ethicon Endo-Surgery, Inc). The remaining gastric tube has an average volume of 80-200 ml. Areas with staple line bleeding are stopped with surgical clips. After methylene blue is injected into the stomach with the help of an orogastric tube and it is confirmed that there is no leakage from the staple line, the previously separated gastrocolic ligament is sutured to the stomach staple line with a v-lock suture. The folds are closed in the anatomical plane.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older and younger than 64 years old.
* At least 5 years of morbid obesity (BMI >40 or >35 comorbidity)
* Patients with temporary or inadequate response (less than 10% of body weight will be considered insufficient) weight loss despite diet for at least 6 months before the operation under the guidance of a dietitian.

Exclusion Criteria:

* Past upper gastrointestinal surgery,
* Paraesophageal (type 2), mixed (type 3), or sliding hiatal hernias of 3 cm or more,
* Patients with esophagitis and/or Barrett's metaplasia in upper gastrointestinal system (GIS) endoscopy
* Those with peripheral vascular disease Those with a history of cerebrovascular accident
* Patients with coagulopathy
* History of chronic analgesic use
* Patients with perioperative complications
* Patients with a previous psychiatric diagnosis other than depression
* Patients who lost less than 10% of their initial weight at the 6th month after the operation
* patients with chronic alcohol use
* patients with recent psychological trauma
* low-income patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing laparoscopic sleeve gastrectomy were included in the study. It was planned to investigate the changes in aggression rates before and after weight loss by applying aggression questionnaires to all patients.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
agression score after weight loss | 1 year
  After significant weight loss in the first year after laparoscopic sleeve gastrectomy, the preoperative aggression questionnaires will be re-administered to all patients.

SECONDARY OUTCOMES:
agression score before weight loss | 1 year
  Aggression questionnaires will be filled in all patients while they are morbidly obese before laparoscopic sleeve gastrectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Study and patient data can be shared upon request.